CLINICAL TRIAL: NCT01781871
Title: Immunogenicity of Repeated Dose 13-valent Pneumococcal Conjugate Vaccine Compared to the Existing Recommended Protocol of Pneumococcal Polysaccharide Vaccine in Adult Kidney and Liver Transplant Patients
Brief Title: Immunogenicity of 13-valent Pneumococcal Conjugate Vaccine Compared to the Pneumococcal Polysaccharide Vaccine in Adult Kidney and Liver Transplant Patients
Acronym: SOT13
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Mari Eriksson, MD, doctor of Infectious Diseases, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HUCH
Record Dates: First submitted 2012-11-22; First posted 2013-02-01 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Kidney Transplantation; Liver Transplantation
Keywords: Pneumococcal vaccination; immunogenicity; solid organ transplant
MeSH Terms: interventions — 13-valent pneumococcal vaccine; Pneumococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Prevenar13 (Experimental): 68 kidney transplant patients vaccinated with Prevenar13 as they enter the transplant waiting list. Pre- and postvaccination serotype specific ELISA and OPA measured. Revaccination at 6 months after the transplantation with Prevenar13, again pre- and postvaccination serotype specific ELISA and OPA measured
  Interventions: Biological: Prevenar13
- Pneumovax (Active Comparator): 68 kidney transplant patients vaccinated with Pneumovax as they enter the transplant waiting list, serotype specific ELISA and OPA measured before and after the vaccination. At six and seven months after transplantation ELISA and OPA measured parallel to the experimental group
  Interventions: Biological: Pneumovax
- liver Prevenar13 (Experimental): 30 liver transplant patients vaccinated with Prevenar13 once they enter the transplant waiting list. Serotype specific ELISA and OPA measured before and after the vaccination. Revaccinated with Prevenar13 at 6 months after the transplantation. ELISa and OPA measured pre- and postvaccination.
  Interventions: Biological: Prevenar13
- liver Pneumovax (Active Comparator): 30 liver transplant patients vaccinated with Pneumovax once they enter the transplant waiting list. Serotype specific ELISA and OPA measured pre- and postvaccination. At 6 and 7 months posttransplant ELISA and OPA measured parallel to the experimental group.
  Interventions: Biological: Pneumovax

INTERVENTIONS:
Biological: Prevenar13 — Prevenar13 0.5ml injected intramuscularly (im.) at day 1 and at 6 months after the transplantation.
  Arms: Prevenar13; liver Prevenar13
Biological: Pneumovax — 0.5ml Pneumovax injected intramuscularly at day 1.
  Arms: Pneumovax; liver Pneumovax

SUMMARY:
Severe Pneumococcal disease, such as bacteremia, meningitis and pneumonia, cause significant morbidity and mortality in both otherwise healthy adult population and in the immunocompromised patients. The incidence rate of invasive pneumococcal disease is considerably higher among organ transplant patients than in healthy individuals. Routine immunization with Pneumococcal vaccine is recommended pretransplant and once 3-5 years after the transplantation. The efficacy and immunogenicity of Pneumococcal polysaccharide vaccine(Pneumovax®) is suboptimal in this patient group. The conjugate Pneumococcal vaccine has been shown to be more immunogenic and safe in some other subgroups of immunocompromised patients. We intend to compare the immunogenicity of repeated dose 13-valent Pneumococcal conjugate vaccine (Prevenar13®)to the existing recommended protocol of Pneumococcal polysaccharide vaccine (Pneumovax®) in adult kidney and liver transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* consecutive new kidney or liver transplantation in our center
* kidney or liver retransplantation in our center

Exclusion Criteria:

* Age < 18 years
* Previous Pneumococcal vaccination < 3 years ago
* Febrile illness at the time of vaccination
* Any sign of graft failure or rejection at the time of vaccination
* Splenectomy
* Pregnancy
* Critically ill patient due to any cause, including terminal uncompensated liver disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2013-01; Primary Completion 2017-10-04 (Actual); Study Completion 2017-10-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline serum serotype specific immunoglobulin G (IgG) antibodies to 13 polysaccharides and their opsonophagocytic activity (OPA) after the first vaccination | baseline and 4 weeks after the first vaccination
Change from baseline serum serotype specific IgG antibodies to 13 polysaccharides and their opsonophagocytic activity (OPA) after the second Prevenar vaccination | baseline and 4 weeks after the second vaccination

SECONDARY OUTCOMES:
vaccination reactions | from vaccination upto 1 week
  Questionaire and phone interview assessment of vaccination reactions and adverse effects.
rejection | at 1 and 2 months after the vaccination
  Urine analyses and creatinine measurement with kidney transplant patients. Alanine aminotransferase measurement with liver transplant patients.

CONTACTS AND LOCATIONS:
Overall Officials: Veli-Jukka Anttila, MD,PhD,Docent, Principal Investigator — HUCH
Locations (2):
- Finland (2):
  - Helsinki University Central Hospital, Helsinki, HUS
  - Heikki Saha, Tampere

IPD SHARING:
Plan to Share IPD: Undecided